CLINICAL TRIAL: NCT00646035
Title: A Phase III, Prospective, Placebo-Controlled, Double-Blind, Randomized, Multi-Center Study to Evaluate the Safety and Efficacy of Paricalcitol Capsules in Reducing Serum Intact Parathyroid Hormone Levels in End Stage Renal Disease Subjects on Peritoneal Dialysis
Brief Title: A Study to Evaluate the Safety and Efficacy of Paricalcitol Capsules in Reducing Serum Intact Parathyroid Hormone Levels in End Stage Renal Disease Subjects on Peritoneal Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Keith Boardway, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001-015; R&D/02/655
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: paricalcitol capsules
- B (Placebo Comparator)
  Interventions: Drug: paricalcitol capsules

INTERVENTIONS:
Drug: paricalcitol capsules — baseline iPTH/60
  Other Names: ABT-358; Zemplar; paricalcitol

SUMMARY:
To determine the safety and efficacy of paricalcitol capsules as compared to placebo for treatment of secondary hyperparathyroidism by decreasing serum intact parathyroid hormone levels in end stage renal disease subjects on peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than or equal to 18 years.
* Subject is diagnosed with ESRD and must be on continuous PD 7 days per week for at least 2 months prior to Screening Phase.
* If female, subject is either not of childbearing potential or is of childbearing potential and practicing one of the recommended methods of birth control.
* If female, subject must have a negative serum pregnancy test prior to treatment.
* If female, subject is not breastfeeding.
* Subject is undergoing full PD regimen and is expected to remain on this PD regimen for the duration of the study.
* For those subjects who have been taking a phosphate binder prior to therapy, the subject has been on a stable type of phosphate binder at least 4 weeks prior to the Pre-Treatment Phase.
* For entry into the Pretreatment Phase the subject must have: Calcium level less than or equal to 10.5 mg/dL and Ca x P level less than or equal to 65.
* For entry into the Treatment Phase the subject must have: iPTH greater than or equal to 300 pg/mL, calcium level of 8.0 to 10.5 mg/dL, inclusive, and Ca x P less than or equal to 65.
* Subject has voluntarily signed and dated an IRB approved informed consent.

Exclusion Criteria:

* Subject has history of an allergic reaction or significant sensitivity to drugs similar to the study drug
* Subject has had active peritonitis within 1 month prior to screening phase.
* Subject has had more than one episode of peritonitis within 4 months prior to screening phase.
* Subject has received a partial parathyroidectomy within 1 year prior to screening phase.
* Subject has had acute renal failure within 3 months of screening phase.
* Subject has chronic gastrointestinal disease.
* Subject has taken aluminum-containing phosphate binders for greater than 3 weeks in the last 3 months prior to the screening phase or will require these medications greater than 3 weeks in the study.
* Subject has a current malignancy or clinically significant liver disease.
* Subject has a history of drug or alcohol abuse within 6 months prior to screening phase.
* Subject has evidence of poor compliance with diet, medication, or PD.
* Subject has participated in any investigational drug or device study within 4 weeks prior to the treatment phase.
* Subject is taking maintenance calcitonin, glucocorticoids, or other drugs that may affect calcium or bone metabolism, other than females on stable estrogen and/or progestin therapy.
* For any reason, subject is considered by the investigator to be an unsuitable candidate to receive paricalcitol capsules.
* Subject is known to be HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2002-01; Primary Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
The achievement of two consecutive greater than or equal to 30% decreases from baseline iPTH levels. | 12 weeks
The incidence of clinically meaningful hypercalcemia and elevated Ca x P. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (22):
- United States (21):
  - Los Angeles, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Fort Myers, Florida
  - Tampa, Florida
  - Savannah, Georgia
  - Evanston, Illinois
  - Maywood, Illinois
  - Indianapolis, Indiana
  - New Orleans, Louisiana
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Mineola, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Lubbock, Texas
- Krakow, Poland